CLINICAL TRIAL: NCT07050446
Title: Multicentre, Randomized, Controlled, Double-blind, Parallel Design Clinical Study to Evaluate the Efficacy, Safety and Tolerability of Vizol S DIGI EYE in the Adult Patient Population With Moderate to Severe Dry Eye Disease for up to 28 Days
Brief Title: Vizol S DIGI EYE Efficacy and Safety Study in Patients With Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jadran Galenski laboratorij d.d. (Industry)
Collaborators: Poseidon Clinical Research Balkans LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: JGL02-Vizol S_DIGI EYE 23
Record Dates: First submitted 2025-06-24; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Dry Eye Disease (DED)
Keywords: KCS; DED; dry eye syndrome; moderate dry eye disease; severe dry eye disease; evaporative DED; menthol; digital device; digital screen; eye strain; fatigue; keratoconjunctivitis sicca (KCS)
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia; Fatigue; Keratoconjunctivitis Sicca | interventions — Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Multicentre, randomized, controlled, double-blind, parallel design clinical study
Who Masked: Participant, Care Provider, Investigator
Masking Description: As the clinical trial will be conducted in a double-blind way, both investigators and patients will be blind with respect to the treatment administered. For the purpose of individual unblinding of a patient's treatment the investigator will receive a sealed emergency envelope for each patient containing the treatment code (Only in case of medical emergency it is permitted to open the emergency envelope).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vizol S DIGI EYE (Experimental): topical administration of 1 drop of Vizol S DIGI EYE in each eye 4 times a day for 28 days
  Interventions: Drug: Vizol S DIGI EYE eye drops
- 0,9% saline solution, eyedrops (Placebo Comparator): topical administration of 1 drop of 0,9% saline solution, eyedrops matching Vizol S DIGI EYE in each eye 4 times a day for 28 days
  Interventions: Drug: 0,9% saline solution, eye drops

INTERVENTIONS:
Drug: Vizol S DIGI EYE eye drops — 1 drop 4 times a day
  Other Names: Test; (T)
  Arms: Vizol S DIGI EYE
Drug: 0,9% saline solution, eye drops — 1 drop 4 times a day
  Other Names: Control; (C)
  Arms: 0,9% saline solution, eyedrops

SUMMARY:
The clinical investigation was intended to investigate the efficacy, ocular tolerability and safety of Vizol S DIGI EYE, a new eye drops, solution developed by JADRAN - GALENSKI LABORATORIJ d.d., in patients with moderate to severe evaporative DED after a treatment for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* Diagnosis of moderate to severe dry eye disease (DED) with a baseline
* Ocular Surface Disease Index (OSDI) score ≥23 (approximately 15% of the population should wear contact lenses);
* Tear Film Break-Up Time (TBUT) <10 s in one or both eyes at baseline;
* National Eye Institute (NEI) score for corneal fluorescein surface staining >5/15 and for conjunctival fluorescein surface staining >6/18 at baseline;
* Best corrected visual acuity (BCVA) of ≥20/80 (or ≥55 letters score or ≥0.6 Early Treatment Diabetic Retinopathy Study log of the minimum angle of resolution value) in both eyes at screening;
* Use of electronic devices (e.g., computers, laptops, smart phones, tablets, televisions (TVs), electronic book readers) with digital screens for more than 6 hours daily;
* Use of eyelid hygiene for at least 14 days prior to screening;
* Written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the patients participating in the clinical trial.

Exclusion Criteria:

* History of hypersensitivity or intolerance to any component of investigational product (IP);
* History of hypersensitivity to fluorescein;
* Any active ocular disease or any anterior ocular surface findings (diseases and irregularities) other than dry eye disease;
* Ocular or refractive surgery (e.g., LASIK, photorefractive keratectomy (PRK) etc.) within the last 12 months from screening;
* Current punctual occlusion of any type;
* History of ocular trauma;
* History of herpes simplex or herpes zoster keratitis;
* History of any type of corneal ulcers;
* Any other acute or chronic disease which may interfere with the aims of the clinical trial or other relevant ocular pathology judged by the investigator that preclude safe administration of the IPs;
* Systemic diseases that alter the ocular surface;
* History of severe allergies or multiple drug allergies unless it is judged as not relevant for the clinical trial by the investigator;
* History of malignancy (other than localized basal cell carcinoma of the skin or in situ cervical cancer);
* Use any topical ophthalmic medication within the last 30 days (except for artificial tears or lubricants; patients will be required to discontinue any other artificial tear or lubricants within the last 14 days and during the trial);
* Use of systemic medications that may contribute to dry eye (unless on a stable regimen for ≥30 days before screening and throughout the study);
* History of or current drug or alcohol dependence;
* Positive Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) test;
* History of Coronavirus Disease 2019 (COVID-19) within the last 30 days (to be defined in line with national requirements);
* History of direct contact with insufficient protection to persons with COVID-19 within the last 14 days (to be defined in line with national requirements);
* Pregnancy or breastfeeding;
* Female patients with childbearing potential (any female after menarche unless postmenopausal for ≥12 months, or surgically sterilized) who are not willing to use a highly effective method of contraception during the study;
* Positive pregnancy test, for female patients with childbearing potential only;
* Patients suspected or known not to follow instructions;
* Patients who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the clinical trial;
* Participation in another clinical trial within 3 months before screening or over a period of 5 half-lives, or double duration of the biological effect of the investigational product received, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Mean change in the tear film break-up time (TFBUT) from Visit 1 (baseline) to Visit 2 (day 14) | baseline and week 2 follow up
  Tear film break-up time (TBUT) will be assessed following the instillation of fluorescein solution into the eye. Fluorescein will be instilled at the outer canthus to avoid ocular surface damage, with the excess saline on the strip shaken off, or a reduced area fluorescein strip used. Viewing will take place between 1 and 3 min after instillation.
  Two measurements per eye will be performed and the mean value documented and used for evaluation.

SECONDARY OUTCOMES:
Mean change in the tear film break-up time (TFBUT) from Visit 1 (baseline) to Visit 3 (day 28) | baseline and week 4 follow up
  Tear film break-up time (TFBUT) will be assessed following the instillation of fluorescein solution into the eye. Fluorescein will be instilled at the outer canthus to avoid ocular surface damage, with the excess saline on the strip shaken off, or a reduced area fluorescein strip used. Viewing will take place between 1 and 3 min after instillation. Two measurements per eye will be performed and the mean value documented and used for evaluation
percent (%) change in the tear film break-up time (TFBUT) from Visit 1 (baseline) to Visit 2 (day 14) and from Visit 1 (baseline) to Visit 3 (day 28) | baseline and week 2 follow-up; baseline and week 4 follow-up
  Tear film break-up time (TFBUT) will be assessed following the instillation of fluorescein solution into the eye. Fluorescein will be instilled at the outer canthus to avoid ocular surface damage, with the excess saline on the strip shaken off, or a reduced area fluorescein strip used. Viewing will take place between 1 and 3 min after instillation. Three measurements per eye will be performed and the mean value documented and used for evaluation
change in the tear film break-up time (TFBUT) on Visit 1 (day 1) | baseline and 4 hour after 1st application
  Tear film break-up time (TBUT) will be assessed following the instillation of fluorescein solution into the eye. On Day 1 TBUT will be assessed at two time points (baseline and 4 hours post-dose). Fluorescein will be instilled at the outer canthus to avoid ocular surface damage, with the excess saline on the strip shaken off, or a reduced area fluorescein strip used. Viewing will take place between 1 and 3 min after instillation.
  Two measurements per eye will be performed and the mean value documented and used for evaluation.
Mean change in ocular surface disease index (OSDI) score from Visit 1 (baseline) to Visit 2 (day 14) and Visit 3 (day 28) | baseline, week 2 follow-up and week 4 follow-up
  Symptoms of DED will be assessed using the Ocular Surface Disease Index (OSDI) questionnaire at each visit. The 12-item OSDI questionnaire scores range from 0 to 100, it contains 3 ocular symptom questions, 6 vision-related function questions, and 3 environmental trigger questions. Each question score ranges from 0 ("none of the time") to 4 ("all of the time"). The total score is calculated based on the following formula: Total score: OSDI = ([sum of scores for all questions answered*100]/[total number of questions answered*4]).
Mean changes in ocular surface staining score (OSS) (total corneal and total conjunctival staining score) from Visit 1 (baseline) to Visit 2 (day 14) and Visit 1 to Visit 3 (day 28) | baseline, week 2 follow-up and week 4 follow-up
  Ocular surface staining of five corneal regions and six conjunctival regions will be observed at each visit by slit-lamp examination after instillation of fluorescein respectively. Surface staining will be scored as 0 (normal, no staining), 1 (mild, superficial stippling or macropunctate staining), 2 (moderate, macropunctate staining with some coalescent areas), or 3 (severe, numerous coalescent macropunctate areas or patches). Scores will be summed to yield total corneal and total conjunctival staining scores for each eye.
Change in Dry Eye Symptom Score (DESS) on Visit 1 (day 1) | baseline and 0, 4 and 8±1 hour after 1st application
  Dry Eye Symptom Score will be assessed, using a 10-point Likert scale, where 0 indicates no symptoms and 10 indicates the most severe symptoms, based on the change from baseline in dry eye symptom scores on day 1 (baseline and 0, 4, and 8±1 hours after 1st dose application). Median values will be documented and used for evaluation.
Change in Soothing Sensation Score (SSS) on Visit 1 (day 1) | baseline and 0, 4 and 8±1 hour after 1st application
  Soothing Sensation Score will be assessed, using a 10-point Likert scale, where 0 indicates no symptoms and 10 indicates the most severe symptoms, based on the change from baseline in soothing sensation scores on day 1 (baseline and 0, 4, and 8±1 hours after 1st dose application). Median values will be documented and used for evaluation.
Change in Refreshing Effect Score (RES) on Visit 1 (day 1) | 0, 0.25 and 1 hour after 1st application
  Refreshing Effect Score will be assessed, using a 10-point Likert scale on day 1 (0, 0.25 and 1 hour after 1st dose application), where 0 indicates no symptoms and 10 indicates the most severe symptoms. Median values will be documented and used for evaluation.

OTHER OUTCOMES:
The presence of Adverse Event/ /Serious Adverse Event (AE/ /SAE) throughout the investigation period | baseline, week 2 follow-up and week 4 follow-up
  The patients will be asked to report any Pre-Treatment Sign and symptom/Adverse Events (PTSS/AEs) spontaneously.
Best-corrected visual acuity (BCVA) | baseline, week 2 follow-up and week 4 follow-up
  Best corrected visual acuity (BCVA) will be assessed at each visit. BCVA assessment will be at 4 meters using an ETDRS chart (The Early Treatment Diabetic Retinopathy Study Group). Results will be calculated as logMAR scores. The logMAR scale (logarithm of the Minimum Angle of Resolution) ranges approximately from -0.3 to 1.0, where lower scores indicate better visual acuity and higher scores indicate worse visual acuity.
Frequency of ocular signs | baseline, week 2 follow-up and week 4 follow-up
  Ocular signs will be assessed by slit-lamp examination at all study visits. The following signs will be assessed: • active inflammation or significant structural change or discharge (eyelids and conjunctiva); • active inflammation or active structural change, including focal scarring and fine deposition (cornea); • active inflammation (iris and anterior chamber); • level of lens opacity, pseudophakia, or aphakia (lens, with an emphasis on the visual axis)
Change in tolerability assessment score (TAS) on Visit 1 (day 1) | Day 1
  Tolerability Assessment Score will be assessed on Day 1 following instillation. The symptoms (burning sensation, stinging sensation, blur, and foreign body sensation) will be evaluated using a a 10-point Likert scale, where 0 indicates no symptom and 10 indicates the most severe symptom. Tolerability Assessment Score will be listed and evaluated descriptively (number of patients (N), arithmetic mean, standard deviation (SD), median, minimum, and maximum). Results for 0-5 and 6-10 scores will be summarized using counts and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: D. Veselinović, Prof. dr, Principal Investigator — Specialized clinic for eye disease - klinika Veselinović
Locations (3):
- Serbia (3):
  - Special eye hospital - Beogradski oftalmološki centar, Belgrade, Belgrade
  - Laser Centre Vid, Kragujevac, Kragujevac
  - Specialized clinic for eye disease - klinika Veselinović, Niš, Niš

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) are available to the Health Authorities upon request

REFERENCES:
- [Background] Novack GD, Asbell P, Barabino S, Bergamini MVW, Ciolino JB, Foulks GN, Goldstein M, Lemp MA, Schrader S, Woods C, Stapleton F. TFOS DEWS II Clinical Trial Design Report. Ocul Surf. 2017 Jul;15(3):629-649. doi: 10.1016/j.jtos.2017.05.009. Epub 2017 Jul 20. PMID 28736344
- [Background] Chiambaretta F, Doan S, Labetoulle M, Rocher N, Fekih LE, Messaoud R, Khairallah M, Baudouin C; HA-trehalose Study Group. A randomized, controlled study of the efficacy and safety of a new eyedrop formulation for moderate to severe dry eye syndrome. Eur J Ophthalmol. 2017 Jan 19;27(1):1-9. doi: 10.5301/ejo.5000836. Epub 2016 Jul 20. PMID 27445067
- [Background] Aguilar AJ, Marquez MI, Albera PA, Tredicce JL, Berra A. Effects of Systane((R)) Balance on noninvasive tear film break-up time in patients with lipid-deficient dry eye. Clin Ophthalmol. 2014 Nov 25;8:2365-72. doi: 10.2147/OPTH.S70623. eCollection 2014. PMID 25473263
- [Background] Wolffsohn JS, Arita R, Chalmers R, Djalilian A, Dogru M, Dumbleton K, Gupta PK, Karpecki P, Lazreg S, Pult H, Sullivan BD, Tomlinson A, Tong L, Villani E, Yoon KC, Jones L, Craig JP. TFOS DEWS II Diagnostic Methodology report. Ocul Surf. 2017 Jul;15(3):539-574. doi: 10.1016/j.jtos.2017.05.001. Epub 2017 Jul 20. PMID 28736342